CLINICAL TRIAL: NCT04271085
Title: Living Well, Dying Well. a Research Programme to Support Living Until the End (iLIVE)
Brief Title: Living Well, Dying Well. a Research Programme to Support Living Until the End
Acronym: iLIVE
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: University of Liverpool (Other); Klinikum der Universität Köln (Other); Lund University (Other); The University Clinic of Pulmonary and Allergic Diseases Golnik (Other); University of Bern (Other); Cudeca Hospice Foundation (Other); Helse-Bergen HF (Other); Landspitali University Hospital (Other); Pallium Latinoamérica N.G.O (Other); University of Humanistic Studies (Unknown); Medical University of Vienna (Other); Arohanui Hospice Service Trust (Unknown)
Responsible Party: Principal Investigator, Agnes van der Heide, Professor, Erasmus Medical Center
Other Study IDs: H2020-825731
Record Dates: First submitted 2019-12-27; First posted 2020-02-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-09

CONDITIONS: Terminal Care
Keywords: Patients in the last phase of life
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients in the last phase of life: Patients in the last phase of life and their families
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention involved

SUMMARY:
The iLIVE project involves a cohort study in which patients with an estimated life expectancy of six months or less are followed until they die. In total, the investigators will include 2200 patients in 11 countries, i.e. 200 per country. The primary outcome for the cohort study is a descriptive assessment of the concerns, expectations and preferences around dying and end-of-life care of patients and their relatives, in different settings and cultures..

DETAILED DESCRIPTION:
Rationale: In the EU about 4 million people yearly die from a chronic illness. Many of these people die in pain or distress. Care for dying patients and their close relatives is often suboptimal.

Objective: To contribute to high-quality personalized care at the end of life by:

1. Providing in-depth understanding of the concerns, expectations and preferences of patients in the last phase of life and their relatives
2. Understanding the cultural, gender, age, healthcare -related and socio-economic variance in these concerns expectations and preferences Study design: The iLIVE project involves a cohort study in which patients with an estimated life expectancy of six months or less are followed until they die. In total, the investigators will include 2200 patients in 11 countries, i.e. 200 per country. Participants are requested to also involve a close relative. Both patients and relatives are asked to fill in a questionnaire, at baseline and after four weeks. If patients die during the study, the relative is asked to fill in a post-bereavement questionnaire. Medical files are studied to assess health care use in the last days of life.

Main study endpoints: The primary outcome for the cohort study is a descriptive assessment of patients' concerns, expectations and preferences around dying and end-of-life care, at baseline and after one month of follow-up.

Potential risks and benefits associated with participation: The study population concerns vulnerable people who may experience fluctuating symptoms and levels of suffering across their disease trajectory. The investigators acknowledge the risk of overburdening or stigmatizing participants. If patients feel burdened by participating in the study, they are encouraged to indicate that. The investigators will develop a protocol for researchers and interviewers to address such situations.

ELIGIBILITY:
Inclusion Criteria patients:

* The patient is aware that recovering from his/her disease is unlikely, to be assessed by the attending physician
* The attending physician would not be surprised if the patient were to die within 6 months
* If the physician is uncertain about the surprise question, the patient is eligible if presenting with at least one SPICT indicator:

General SPICT indicators:

* Unplanned hospital admission
* Performance status is poor or deteriorating, with limited reversibility (eg stays in bed or in a chair for more than half the day)
* Depends on others for care due to increasing physical and/or mental health problems; person's carer needs more help and support
* Progressive weight loss; remains underweight; low muscle mass
* Persistent symptoms despite optimal treatment of underlying condition(s)
* Person (or family) asks for palliative care; chooses to reduce, stop or not have treatment; or wishes to focus on quality of life

Disease-specific SPICT indicators:

Cancer:

* Functional ability deteriorating due to progressive cancer
* Too frail for cancer treatment or treatment is for symptom control

Neurological disease:

* Progressive deterioration in physical and/or cognitive function despite optimal therapy
* Speech problems with increasing difficulty communicating and/or progressive difficulty with swallowing
* Recurrent aspiration pneumonia; breathless or respiratory failure
* Persistent paralysis after stroke with significant loss of function and ongoing disability

Heart/vascular disease:

* Heart failure or extensive, untreatable coronary artery disease; with breathlessness or chest pain at rest or on minimal effort
* Severe, inoperable peripheral vascular disease

Respiratory disease:

* Severe, chronic lung disease; with breathlessness at rest or on minimal effort between exacerbations
* Persistent hypoxia needing long term oxygen therapy
* Has needed ventilation for respiratory failure or ventilation is contraindicated

Kidney disease:

* Stage 4 or 5 chronic kidney disease (eGFR < 30ml/min) with deteriorating health
* Kidney failure complicating other life limiting conditions or treatments
* Stopping or not starting dialysis

Liver disease:

* Cirrhosis with one or more complications in the past year: diuretic resistant ascites; hepatic encephalopathy; hepatorenal syndrome; bacterial peritonitis; or recurrent variceal bleeds
* Liver transplant is not possible

Dementia/ frailty:

* Unable to dress, walk or eat without help
* Eating and drinking less, difficulty with swallowing
* Urinary and faecal incontinence
* Not able to communicate by speaking; little social interaction
* Frequent falls; fractured femur
* Recurrent febrile episodes or infections, aspiration pneumonia

Other conditions:

o Deteriorating and at risk of dying with other conditions or complications that are not reversible; any treatment available will have a poor outcome

Exclusion Criteria patients:

* The patient is incapable of filling in a questionnaire in the country's main language or in English (patients may be supported by relatives when filling in the questionnaire)
* The patient is incapable of providing informed consent to participate in the study, to be assessed by the attending physician

Inclusion Criteria relatives:

* Family, friend or other close relative of the patient
* 18 years or older
* The relative is aware that it is unlikely that that patient will recover from his/her disease

Exclusion Criteria relatives:

* The relative is incapable of filling in a questionnaire in the country's main language or in English
* The relative is incapable of providing informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All competent adult patients with an estimated life expectancy of six months or less are eligible, regardless of their diagnosis, gender or age, or place of residence, and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Concerns, expectations and preferences around dying and end-of-life care (descriptive assessment of prevalence) | Baseline
  Self developed questions, adapted from the Serious Illness Conversation Guide and the AEOLI questionnaire.
Concerns, expectations and preferences around dying and end-of-life care (descriptive assessment of prevalence) | One month of follow-up
  Self developed questions, which were inspired by the Serious Illness Conversation Guide and the AEOLI questionnaire.

SECONDARY OUTCOMES:
Edmonton Symptom Assessment Scale (range 0-10, with higher score meaning worse outcome) | At baseline and after one month of follow-up
  Symptoms
European Organisation for Research and Treatment of Cancer Quality of Life C15-Palliative Care questionnaire, quality of life item (range 1-7, with higher score indicating better outcome) | At baseline and after one month of follow-up
  Quality of life
EuroQol-5d questionnaire (range 1-5 per item, with higher score indicating worse outcome) | At baseline and after one month of follow-up
  Quality of life
ICECAP Supportive Care Measure (range 1-4 per item, with higher score indicating worse outcome) | At baseline and after one month of follow-up
  Experience of support
Use of medical interventions (hospitalisation, medication, surgery, other interventions) | One week
  Retrospective assessment for patients who die during follow-up of medical interventions in the last week of patients' life, using a self-developed checklist
Bereaved relatives' experiences | 8-10 weeks post-bereavement
  International Care of the dying questionnaire (descriptive), Hogan Grief Reaction Checklist (despair (13 items) and personal growth (12 items) scales, range 1-5 per item)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes van der Heide, PhD, Principal Investigator — Erasmus Medical Center
Locations (11):
- Pallium Latinoamérica, Buenos Aires, Argentina
- University Hospital Cologne, Cologne, Germany
- Landspitali National University Hospital of Iceland, Reykjavik, Iceland
- Agnes van der Heide, Rotterdam, Netherlands
- Arohanui Hospice Service, Palmerston North, New Zealand
- Haukeland University Hospital, Bergen, Norway
- University Clinic for Respiratory and Allergic Diseases Golnik, Ljubljana, Slovenia
- Centro de Cuidados Paliativos Cudeca, Málaga, Spain
- Skåne University Hospital, Lund, Sweden
- Bern University Hospital, Bern, Switzerland
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided